CLINICAL TRIAL: NCT02698085
Title: Effectiveness of Physiotherapy Treatment With Diacuteneous Fibrolysis in Patients With Carpal Tunnel Syndrome
Brief Title: Diacutaneous Fibrolysis on Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Sandra Jiménez, Principal investigator, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C.I.PI14/00086
Record Dates: First submitted 2016-02-03; First posted 2016-03-03 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Carpal Tunnel Syndrome
Keywords: carpal tunnel syndrome; physiotherapy; manual therapy
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Goup (Experimental): Actual Diacutaneous Fibrolysis
  Interventions: Other: Actual Diacutaneous Fibrolysis
- Placebo Group (Sham Comparator): Sham Diacutaneous Fibrolysis
  Interventions: Other: Sham Diacutaneous Fibrolysis

INTERVENTIONS:
Other: Actual Diacutaneous Fibrolysis — Diacutaneous Fibrolysis is a non invasive physiotherapeutic technique applied by means of a set of metallic hooks ending a spatula with bevelled edges that help to treat the muscles and conjunctive tissues and trying to improve mobility between mobility between muscle planes.
  Arms: Intervention Goup
Other: Sham Diacutaneous Fibrolysis — Sham Diacutaneous Fibrolysis is applied at a superficial level. A pinch of skin was held with the thumb of the palpatory hand and the tip of the spatula but without effect in the muscle because no penetrate in deep tissue
  Arms: Placebo Group

SUMMARY:
Diacutaneous Fibrolysis is a manual method of treatment, addressed to mechanical pain of the neuromusculoskeletal system. In the clinical practice a favorable effect is observed in patients with carpal tunnel syndrome, but there is no published studies evaluating the results os this technique.

The objective of this trial is to evaluate if Diacutaneous Fibrolysis is more effective in symptoms, function, grip, mechanosensitivity and neural conduction velocity compared to a placebo.

For this purpose the investigators conduct a randomized controlled trial double-blind (patient and examiner). The investigators included patients diagnosed of carpal tunnel syndrome (low to moderate intensity) with a neurophysiological test.

Patients included are randomized into 2 groups one receive Diacutaneous Fibrolysis and the other placebo. Both groups receive 5 treatment sessions.

The variables are measured at the beginning and end of treatment. And also some variables are measured before and after each session. Patients who participated in placebo group, when the intervention finish the investigators will be given the opportunity to receive the actual technique

DETAILED DESCRIPTION:
The investigators selected patients diagnosed with carpal tunnel syndrome with electroneurogram, if they meet the inclusion criteria are offered to take part in this study.

When the patient agree to participate and signed informed consent, the investigators collected dependent variables considered (symptoms, mechanosensitivity, functional capacity with upper limb, tractor speed of neural conduction ...) and the patient is assigned to an intervention group: real or placebo. Each patient receives treatment 5 sessions trascurriendo intersessional 2- 5 days. After 5 sessions the investigators remeasured the same variables. In addition, a month later they remeasured again symptoms and functional capacity with upper limb. Finally, they were shown the technique they have received. If the patient has received the technical placebo he/she is given the opportunity to receive 5 sessions of the actual technique.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed medically with neurophysiological test of carpal tunnel syndrome (low and moderate intensity)

Exclusion Criteria:

* Severe carpal tunnel syndrome
* Previous surgery on the hand
* hormonal factors: diabetes, thyroids pathologies, pregnant
* cervical disfunctions
* ulcerations or skins disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04-01; Primary Completion 2016-09-01 (Actual); Study Completion 2016-10-10 (Actual)

PRIMARY OUTCOMES:
Intensity symptoms pre-intervention with a visual analogic scale | pre-intervention
  The investigators measure the intensity of symptoms with a visual analogic scale at baseline.
Intensity symptoms post-intervention with a visual analogic scale | post-intervention
  The investigators measure the intensity of symptoms with a visual analogic scale at the end of the intervention (2 weeks after pre-intervention) the investigators measured the intensity of symptoms (through study completion, an average 15 days)
Intensity symptoms after month with a visual analogic scale | after month
  The investigators measure the intensity of symptoms with a visual analogic scale after month of post-intervention.

SECONDARY OUTCOMES:
Upper limb function pre-intervention with a validated questionnaire (DASH) | pre-intervention
  The investigators measure upper limb function with a validated questionnaire (DASH), at baseline.
Mechanosensitivity of median nerve pre-intervention with neurodynamic test | Pre-intervention
  The investigators measure the mechanosensitivity of median nerve with neurodynamic test at baseline.
Mechanosensitivity of median nerve post-intervention with neurodynamic test | post-intervention
  The investigators measure the mechanosensitivity of median nerve with neurodynamic test at the end of the intervention (through study completion, an average 15 days).
Neurophysiological test pre-intervention | pre-intervention
  The investigators measure the neurophysiological properties of median nerve with electroneurogram with the neural conduction velocity at baseline
Neurophysiological test post-intervention | post-intervention
  The investigators measure the neurophysiological properties of median nerve with electroneurogram with the neural conduction velocity at the end of the intervention (through study completion, an average 15 days)
Upper limb function post-intervention with a validated questionnaire (DASH) | post-intervention
  The investigators measure upper limb function with a validated questionnaire (DASH) at the end of the intervention (through study completion, an average 15 days)
Upper limb function after month with a validated questionnaire (DASH) | after month
  The investigators measure upper limb function with a validated questionnaire (DASH) after a month post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Sand J, Graduated, Principal Investigator — I
Locations (1):
- Sandra Jiménez, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No
The patient data were confidential and were assigned a number to each patient to maintain confidentiality